CLINICAL TRIAL: NCT02279589
Title: Open Randomized Trial Evaluating Four Anti-pneumococcal Vaccine Strategies With Fractionated Doses of Non Conjugate Polysaccharide Vaccine to Prevent Hyporesponse in Healthy Volunteers
Acronym: HYPOPNEUMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P130903
Record Dates: First submitted 2014-10-16; First posted 2014-10-31 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Pneumococcal Infection
Keywords: hyporesponsiveness; vaccination; recommendations; improvement; schedule; fractional dose; conjugate polysaccharide vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): Description :
  15 subjects with : Prevenar13® 0,5 then Pneumo 23® 0,5 then Pneumo 23® 0,1
  Route : Intramuscular vaccination schedule : M0, M2, M12
  Interventions: Biological: Pneumo 23® 0,5; Biological: Pneumo 23® 0,1; Biological: Prevenar13® 0,5
- Group B (Active Comparator): Description 15 subjects with : Prevenar13® 0,5 then Pneumo 23® 0,1 then Pneumo 23® 0,1
  Route : Intramuscular vaccination schedule : M0, M2, M12
  Interventions: Biological: Pneumo 23® 0,1; Biological: Prevenar13® 0,5
- Group C (Active Comparator): Description :
  15 subjects with : Prevenar13® 0,5 then Pneumo 23® 0,1 then Pneumo 23® 0,5
  Route : Intramuscular vaccination schedule : M0, M2, M12
  Interventions: Biological: Pneumo 23® 0,5; Biological: Pneumo 23® 0,1; Biological: Prevenar13® 0,5
- Group D (Active Comparator): Description:
  15 subjects with : Prevenar13® 0,5 then Pneumo 23® 0,5 then Pneumo 23® 0,5
  Route : Intramuscular vaccination schedule : M0, M2, M12
  Interventions: Biological: Pneumo 23® 0,5; Biological: Prevenar13® 0,5

INTERVENTIONS:
Biological: Pneumo 23® 0,5 — Polysaccharide vaccine Pneumo 23® (Sanofi Pasteur MSD), containing 23 valencies Pneumococcus (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, 33F) administered by intramuscular route. (Deltoid) at full dose. One dose contains: 0, 5 mL of 25 μg of polysaccharide of the 23 serotypes pneumococcus.
  Arms: Group A; Group C; Group D
Biological: Pneumo 23® 0,1 — Polysaccharide vaccine Pneumo 23® (Sanofi Pasteur MSD), containing 23 valencies Pneumococcus (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, 33F) administered by intramuscular route. (Deltoid) at a 1/5 of the dose. One dose contains: 0, 5 mL of 25 μg of polysaccharide of the 23 serotypes pneumococcus.
  Arms: Group A; Group B; Group C
Biological: Prevenar13® 0,5 — The conjugate vaccine Prevenar13® (Pfizer) containing 13 valencies Pneumoccocus (4, 6B, 9V, 14, 18C, 19F, 23F), conjugated with diphtheria anatoxin (CRM 197) administered by intramuscular route (deltoid).
  One dose contains: 0, 5 ml of 2 - 4μg of polysaccharide of the13 serotypes pneumococcus which 12 are shared with Pneumo 23® vaccine conjugated to diphtheria toxoid (CRM 197).

SUMMARY:
Immune response analysis after the combination of PCV13 and PPV23 will lead to evaluate if a prime with PCV13 help to obtain a good response to repeated dose of PPV23.The hyporesponsiveness following the unconjugated vaccine is associated with high polysaccharide antigen concentration. Several issues limit the development and recommendation of anti-pneumococcal vaccine in adult's patients at risk. Reduced doses of unconjugated polysaccharide antigens would bypass the hyporesponsiveness and maintain the expanded coverage serotype.

A better knowledge of immune response following the combination of two vaccines in adults is essential. In addition, adults are required to be exposed to repeated doses of polysaccharide antigens by vaccine or by natural exposure, it is important to determine the extend and duration of any hyporesponsiveness.

The main objective is to evaluate if non conjugate polysaccharidique fractionated doses administered after a conjugate vaccine help to avoid hyporesponse in a schedule with repeated injections of pneumococcal polysaccharidique vaccine

DETAILED DESCRIPTION:
Immune response analysis after the combination of PCV13 and PPV23 will lead to evaluate if a prime with PCV13 help to obtain a good response to repeated dose of PPV23.The hyporesponsiveness following the unconjugated vaccine is associated with high polysaccharide antigen concentration. Several issues limit the development and recommendation of anti-pneumococcal vaccine in adult's patients at risk. Reduced doses of unconjugated polysaccharide antigens would bypass the hyporesponsiveness and maintain the expanded coverage serotype.

A better knowledge of immune response following the combination of two vaccines in adults is essential. In addition, adults are required to be exposed to repeated doses of polysaccharide antigens by vaccine or by natural exposure, it is important to determine the extend and duration of any hyporesponsiveness.

The main objective is to evaluate if non conjugate polysaccharidique fractionated doses administered after a conjugate vaccine help to avoid hyporesponse in a schedule with repeated injections of pneumococcal polysaccharidique vaccine

The projects aims are :

- Primary is to evaluate if non conjugate polysaccharidique fractionated doses administered after a conjugate vaccine help to avoid hyporesponse in a schedule with repeated injections of pneumococcal polysaccharidique vaccine.

Secondary objectives are :

* To study the immune response involved when combining conjugate vaccine (PCV13) and non-conjugate polysaccharide vaccine (PPV23 full dose or fractionated booster dose) and assesses an eventual prime-boost effect.
* To study the impact of fractioned PPV23 on the immune response to PPV23 serotypes, measured as the extension of the serotype coverage.
* To assess the sustainability and evolution of the immune response over time
* To investigate the clinical tolerance to an initial dose of PCV13 followed by repeated doses of PPV23 vaccines
* To describe any invasive infections pneumococcal and community acquired pneumonia occurring during the time course of the study.

Study duration Recruitment: 6 months Participation: 36 months Total duration of the study: 42 month

Study Design Vaccine trial Open randomized 1:1:1:1 phase II comparing the immunogenicity of four pneumococcal vaccination strategies administered by intramuscular route in healthy volunteer's adults aged 18 to 49 years.

Four dose combination of two vaccines will be assessed, Pneumo23® and Prevenar13®. Volunteers will receive three vaccine injections during the study.

Sixty (60) healthy volunteers will be enrolled and randomized into the four following groups:

* Group A: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 one dose of Pneumo23® and at M12, 1/5 dose of Pneumo23®
* Group B: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 1/5 dose of Pneumo23® and at M12, 1/5 dose of Pneumo23®
* Group C: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 1/5 dose of Pneumo23® and at M12, one dose of Pneumo23®
* Group D: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 one dose of Pneumo23® and at M12, one dose of Pneumo23®

Number of visits per volunteer: 9 visits

* 3 vaccination visits: M0, M2, M12
* 6 follow-up visits: M1, M3, M13, M18, M24, M36.
* Unscheduled visit if suspected invasive pneumococcal infection (meningitis, bacteraemia, pneumonia, pleural-pneumonia)

Total number of scheduled subjects :

60 healthy volunteers will be recruited at the CIC 1417: 15 volunteers per group There was no statistical determination of sample size. Data from this trial will identify one or more vaccine strategies that could be tested in clinical trials on population at risk for invasive pneumococcal diseases.

Data from published studies don't give homogeneous references about geometric means titers in OPA with fractional of polysaccharidique vaccine. This is the first study evaluating combined vaccination strategies with a schedule with one initial dose of PCV13 and complete or fractional doses of PPV23.

Expected patient or public health benefit A better assessment of the immunogenicity induced by the combination of Prevenar13® and Pneumo23® will allow to adapt pneumococcal vaccine recommendations for adults. The Pneumo23® has been for a long time the only vaccine recommended in adults with a condition that places them at high risk of invasive pneumococcal infection: splenectomy or functional asplenia, homozygous sickle cell disease, HIV infection (regardless of the immunovirological status), nephrotic syndrome, respiratory failure, heart failure, patients with chronic liver disease, with a history of pulmonary infection or invasive pneumococcal disease. It has to be repeated every 5 years (BEH-vaccination schedule and vaccine recommendations), given the absence of an immune memory. But its immunogenicity is limited and repeated doses may induce hyporesponsiveness. The recent availability of Prevenar13®, polysaccharide conjugate vaccine, in adults led to reassess recommendations for adults advising the combination of two vaccines: PCV13 and PPV23 2 months apart (then repeated doses of PPV23 at 5 years), to induce a response called "prime-boost", that is to say PPV23stimulation of memory response initiated by PCV13 (Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Adults Aged 19 Years and Older - United States, 2013 --MMWR/January 28 2013/Vol. 62). These recommendations need to rely on more solid immunological substrate, including more data in adults whose immune status differs from children. To our knowledge, there is no data examining the various mechanisms of the immune response in the combination of these two vaccines, and taking into account the effect of dose of polysaccharide antigens in the same study, with such immunological monitoring in adults. Data from this clinical trial will therefore support these recommendations, either on the induction of immunological memory response by the PCV13, or on the impact of repeated doses of PPV23. Preventing pneumococcal infections would decrease morbidity; extend life expectancy and quality of life in patients at risk. In a public health perspective, by reducing the number and duration of hospitalization, it would reduce dramatically the vaccine cost.

Study duration Recruitment: 6 months Participation: 36 months Total duration of the study: 42 month

Study Design Vaccine trial Open randomized 1:1:1:1 phase II comparing the immunogenicity of four pneumococcal vaccination strategies administered by intramuscular route in healthy volunteer's adults aged 18 to 49 years.

Four dose combination of two vaccines will be assessed, Pneumo23® and Prevenar13®. Volunteers will receive three vaccine injections during the study.

Sixty (60) healthy volunteers will be enrolled and randomized into the four following groups:

* Group A: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 one dose of Pneumo23® and at M12, 1/5 dose of Pneumo23®
* Group B: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 1/5 dose of Pneumo23® and at M12, 1/5 dose of Pneumo23®
* Group C: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 1/5 dose of Pneumo23® and at M12, one dose of Pneumo23®
* Group D: 15 subjects receiving at M0 one dose of Prevenar13®, at M2 one dose of Pneumo23® and at M12, one dose of Pneumo23®

Number of visits per volunteer: 9 visits

* 3 vaccination visits: M0, M2, M12
* 6 follow-up visits: M1, M3, M13, M18, M24, M36.
* Unscheduled visit if suspected invasive pneumococcal infection

Total number of scheduled subjects :

60 healthy volunteers will be recruited at the CIC 1417: 15 volunteers per group There was no statistical determination of sample size. Data from this trial will identify one or more vaccine strategies that could be tested in clinical trials on population at risk for invasive pneumococcal diseases.

Data from published studies don't give homogeneous references about geometric means titers in OPA with fractional of polysaccharidic vaccine. This is the first study evaluating combined vaccination strategies with a schedule with one initial dose of PCV13 and complete or fractional doses of PPV23.

Expected patient or public health benefit A better assessment of the immunogenicity induced by the combination of Prevenar13® and Pneumo23® will allow to adapt pneumococcal vaccine recommendations for adults. The Pneumo23® has been for a long time the only vaccine recommended in adults with a condition that places them at high risk of invasive pneumococcal infection: splenectomy or functional asplenia, homozygous sickle cell disease, HIV infection (regardless of the immunovirological status), nephrotic syndrome, respiratory failure, heart failure, patients with chronic liver disease, with a history of pulmonary infection or invasive pneumococcal disease. It has to be repeated every 5 years (BEH-vaccination schedule and vaccine recommendations), given the absence of an immune memory. But its immunogenicity is limited and repeated doses may induce hyporesponsiveness. The recent availability of Prevenar13®, polysaccharide conjugate vaccine, in adults led to reassess recommendations for adults advising the combination of two vaccines: PCV13 and PPV23 2 months apart (then repeated doses of PPV23 at 5 years), to induce a response called "prime-boost", that is to say PPV23stimulation of memory response initiated by PCV13 (Advisory Committee on Immunization Practices (ACIP) Recommended Immunization Schedule for Adults Aged 19 Years and Older - United States, 2013 --MMWR/January 28 2013/Vol. 62). These recommendations need to rely on more solid immunological substrate, including more data in adults whose immune status differs from children. To our knowledge, there is no data examining the various mechanisms of the immune response in the combination of these two vaccines, and taking into account the effect of dose of polysaccharide antigens in the same study, with such immunological monitoring in adults. Data from this clinical trial will therefore support these recommendations, either on the induction of immunological memory response by the PCV13, or on the impact of repeated doses of PPV23. Preventing pneumococcal infections would decrease morbidity; extend life expectancy and quality of life in patients at risk. In a public health perspective, by reducing the number and duration of hospitalization, it would reduce dramatically the vaccine cost.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (males and females) of age ≥ 18 to ≤ 49 years old;
* Individuals, who, after the nature of the study have been explained to them, have given written consent according to local regulatory requirements.
* Individuals in good health as determined by the outcome of medical history, physical examination clinical judgement of the investigator.
* Women of childbearing potential must have a negative pregnancy test and an effective contraception during the first 13 months of the study;
* Individuals able to participate and to follow up during the 36 months of the study
* Individuals covered by social security regimen

Exclusion Criteria:

* Individuals with behavioural or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
* Individuals with indication to anti-pneumococcal vaccination at the time of enrolment according to the French vaccination schedule (vaccinal calender BEHn°14-15/2013);
* Individuals with history of pneumococcal vaccination;
* Individuals with history of suspected or low documented invasive pneumococcal infection within the year before enrolment;
* Individuals who have received any another vaccines within 4 weeks prior to enrolment or who are planning to receive any vaccine within the first 13 months of the study; (except Annual influenza vaccination which is permitted 4 weeks before and after each vaccination visit of the study and then allowed at any time during the study follow up)
* Individuals who have received blood, blood products, and/or plasma derivatives including parenteral immunoglobulin preparations in the past 12 weeks before enrolment
* Individuals who have received systemic antibiotic within 7 days before inclusion (except 14 days concerning azithromycine), regardless the duration or dosage
* Individuals with body temperature ≥ 38.0 degrees Celsius within 3 days of study vaccination.
* Individuals with personal or familial history of any illness that, in the opinion of the investigator, might pose additional risk to the subjects due to participation in the study.
* Individual with personal or familial (first degree relatives) history of an auto-immune disorder, or any other known or suspected impairment /alteration of the immune system or under immunosuppressive therapy, including use of systemic corticosteroids (i.e. prednisone, or equivalent) ≥ 10mg/day more than 6 days within the previous 28 days or within 3 days regardless dosage and duration, or in chemotherapy treatment or other immunosuppressive or immunomodulating therapy within the past 168 days (6 months). Topical or inhaled uses of steroid including intranasal are allowed.
* Individuals with thrombocytopenia or coagulation disorder contra-indicating intramuscularly injections; coagulation disorder contra-indicating intramuscularly injections;
* Individuals with evolutionary cancer, cirrhosis, known infection to HIV/ HBV/ HCV or any serious chronic or progressive disease according to the judgment of the investigator
* Individuals with acute respiratory tract infection within the month before enrolment;
* Individuals with history of known allergies/hypersensitivity to any component of both study vaccines;
* Women, who are pregnant or breast-feeding
* Individuals under a measure of legal protection or unable to consent.
* Individuals participating in any clinical trial 28 days prior to first study visit until the M24 visit of the study (+ the day of M36 visit).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Geometric mean antibody titers measured by OpsonoPhagocytose Assay (OPA) at 13 months | 13 months
  The primary end point is the geometric mean antibody titers measured by OPA (OpsonoPhagocytose Assay) for 9 common serotypes to both PPV23 and PCV13 (3, 6B, 7F, 9V, 14,18C, 19A, 19F, 23F), at 1 month after the third dose of vaccine (at M13)

SECONDARY OUTCOMES:
Immune response at 13 months | 13 months
  The immune response involved when combining conjugate vaccine (PCV13) and non-conjugate polysaccharide vaccine (PPV23) and an eventual prime-boost effect will be evaluated by:
  * ELISA antibody concentration against nine common serotypes (3, 6B, 9V, 14,18C, 19A, 19F, 23F, 7F) at month 0, month 1, month 3 and month 13 and proportion of positive serotypes
  * OPA titers against 9 common serotypes (3, 6B, 9V, 14,18C, 19A, 19F, 23F, 7F) at M0, M1, M3 and proportion of positive serotype
  * Measurement of IgG subtypes, measurement of lymphocyte cell phenotypes (memory and naives B cells, marginal zone B cells, follicular zone B cells, B1b and B1a cells), at M0, M1, M3 and M13
Immune response evaluated by ELISA antibody concentration at 36 months | 36 months
  The immune response will be evaluated by ELISA antibody concentration, against 3 uncommon specific serotypes of PPV23 (12F/10A/15B) at M0, M1, M3, M12, M13, M18, M24, M36 and the proportion of positive serotypes (impact of fractionated PPV23)
Sustainability and evolution of the immune response at 36 months | 36 months
  The sustainability and evolution of the immune response over time will be measured by ELISA concentration and OPA titres at regular intervals (M0, M12, M18, M24, and M36) for the 9 PCV13 serotypes to measure changes over time in the immune response.
Clinical tolerance at 36 months | 36 months
  * For 7 days following each vaccination
    • local and/or systemic solicited reactions : Proportion of participants with an event; number, nature, grade and time of occurrence.
  * During the study :
    * Any event related or possibly related to vaccine immunisation: proportion of participant with an event; number, nature, grade and time of occurrence.
    * Any event related to vaccine immunisation and leading to discontinuation of the immunisation regimen: proportion of participant with an event; number, nature, grade and time of occurrence.
    * Serious adverse event, regardless of the relationship to vaccine immunisation: proportion number, nature, grade and time of occurrence
Description of any invasive infections pneumococcal and community acquired pneumonia occurring during 36 months of follow-up | 36 months
  The description of any invasive infections pneumococcal and community acquired pneumonia occurring during the time course of the study will be evaluated by the documentation of invasive bacterial infections with biological and radiological examinations in case of suspected invasive infection (clinical effectiveness)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BODILIS, Principal Investigator — Assistance Publique - Hôpitaux de Paris

REFERENCES:
- [Background] de Roux A, Schmole-Thoma B, Siber GR, Hackell JG, Kuhnke A, Ahlers N, Baker SA, Razmpour A, Emini EA, Fernsten PD, Gruber WC, Lockhart S, Burkhardt O, Welte T, Lode HM. Comparison of pneumococcal conjugate polysaccharide and free polysaccharide vaccines in elderly adults: conjugate vaccine elicits improved antibacterial immune responses and immunological memory. Clin Infect Dis. 2008 Apr 1;46(7):1015-23. doi: 10.1086/529142. PMID 18444818
- [Background] O'Brien KL, Hochman M, Goldblatt D. Combined schedules of pneumococcal conjugate and polysaccharide vaccines: is hyporesponsiveness an issue? Lancet Infect Dis. 2007 Sep;7(9):597-606. doi: 10.1016/S1473-3099(07)70210-4. PMID 17714673
- [Background] Poolman J, Borrow R. Hyporesponsiveness and its clinical implications after vaccination with polysaccharide or glycoconjugate vaccines. Expert Rev Vaccines. 2011 Mar;10(3):307-22. doi: 10.1586/erv.11.8. PMID 21434799
- [Background] Russell FM, Carapetis JR, Balloch A, Licciardi PV, Jenney AW, Tikoduadua L, Waqatakirewa L, Pryor J, Nelson J, Byrnes GB, Cheung YB, Tang ML, Mulholland EK. Hyporesponsiveness to re-challenge dose following pneumococcal polysaccharide vaccine at 12 months of age, a randomized controlled trial. Vaccine. 2010 Apr 26;28(19):3341-9. doi: 10.1016/j.vaccine.2010.02.087. Epub 2010 Mar 4. PMID 20206670
- [Background] Ahman H, Kayhty H, Vuorela A, Leroy O, Eskola J. Dose dependency of antibody response in infants and children to pneumococcal polysaccharides conjugated to tetanus toxoid. Vaccine. 1999 Jun 4;17(20-21):2726-32. doi: 10.1016/s0264-410x(99)00048-1. PMID 10418924